CLINICAL TRIAL: NCT03406962
Title: A Phase 2, Single-arm, Open-label Study to Evaluate the Safety and Efficacy of MGTA-456 in Patients With Inherited Metabolic Disorders (IMD) Undergoing Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: MGTA-456 in Patients With Inherited Metabolic Disorders Undergoing Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Magenta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMD-001
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2020-06

CONDITIONS: Inherited Metabolic Disorders (IMD)
Keywords: inherited metabolic disorders; cerebral adrenoleukodystrophy; Hurler syndrome; globoid cell leukodystrophy; Krabbe disease; metachromatic leukodystrophy; hematopoietic stem cells; hematopoietic stem cell transplant; umbilical cord blood; umbilical cord blood transplant; MGTA-456; myeloablative conditioning regimen; bone marrow transplant; mucopolysaccharidosis-1H
MeSH Terms: conditions — Mucopolysaccharidosis I; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MGTA-456 (Experimental): MGTA-456 is an expanded CD34+ cell therapy investigational product used in replacement of single umbilical cord blood transplantation.
  Interventions: Drug: MGTA-456

INTERVENTIONS:
Drug: MGTA-456 — Hematopoietic stem cell transplantation will be done with the cell therapy product MGTA-456.
  Other Names: HSC835

SUMMARY:
This study is designed to assess the safety and efficacy of using MGTA-456 in patients with Inherited Metabolic Disorders (IMD) undergoing stem cell transplantation.

DETAILED DESCRIPTION:
This phase 2 study is designed to evaluate the safety and efficacy of MGTA-456 in patients with IMD after receiving myeloablative conditioning and HSCT. MGTA-456 is an expanded CD34+ cell therapy product candidate given to induce rapid and sustained hematopoietic engraftment. In patients with selected IMDs, transplant is expected to replace defective or missing protein and preserve neurodevelopment. Since MGTA-456 offers increased numbers of HSCs over standard umbilical cord blood, it is expected to reduce the risks of prolonged neutropenia and thrombocytopenia and graft failure, and potentially transplant-related mortality (TRM). Patients with Hurler syndrome (also referred to as mucopolysaccharidosis-1H (MPS-1H)), cerebral adrenoleukodystrophy (cALD), metachromatic leukodystrophy (MLD) or globoid cell leukodystrophy (GLD) (also referred to as Krabbe disease) are eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age < 2.5 years with Hurler syndrome, age 2-17 years with cerebral adrenoleukodystrophy (cALD), age < 16 years with metachromatic leukodystrophy (MLD) and age ≤ 10 years with globoid cell leukodystrophy (GLD) (also referred to as Krabbe)
* Cord blood grafts require genetic testing and/or demonstration of enzyme activity for patients with Hurler syndrome, MLD or GLD and are tested for very long chain fatty acids (VLCFA) to confirm there is no evidence of VLCFA consistent with ALD
* Adequate organ function
* Availability of eligible donor material

Exclusion Criteria:

* Availability of a matched-related donor who is not a carrier of the same genetic defect
* Active infection at screening
* Prior myeloablative conditioning
* History of human immunodeficiency virus (HIV) infection

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magenta Study Coordinator, Study Director — Magenta Therapeutics
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were referred to clinical sites.
Pre-assignment Details: Before an enrolled patient was infused with MGTA-456, the patient had to undergo a protocol-defined conditioning regimen and the proper expansion and manufacture of MGTA-456 investigational cell therapy product was confirmed.
Period: Overall Study
Arm/Group | MGTA-456
Started | 8
Completed | 5
Not Completed | 3
Not completed — Death | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | MGTA-456
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.49 (2.765)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Height [Mean (Standard Deviation); unit: cm] | 84.44 (23.419)
Weight [Mean (Standard Deviation); unit: kg] | 13.74 (7.863)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment
Description: Engraftment is defined as achieving an absolute neutrophil count (ANC) ≥0.5 × 10⁹/L for 3 consecutive days.
Time Frame: 42 days
Population: Patients who received MGTA-456 investigational product
Measure: Count of Participants; unit: Participants
Groups:
- MGTA-456 Cohort 1: Patients receiving freshly-prepared MGTA-456 CD34+ cell therapy investigational product in replacement of single umbilical cord blood transplantation
- MGTA-456 Cohort 2: Patients receiving cryopreserved MGTA-456 CD34+ cell therapy investigational product in replacement of single umbilical cord blood transplantation
Arm/Group | MGTA-456 Cohort 1 | MGTA-456 Cohort 2
Number analyzed (Participants) | 6 | 2
Participants | 6 | 2

2. Secondary Outcome: Number of Participants With Infusion Toxicities
Description: Incidence of treatment-emergent adverse events (AEs) within 48 hours after MGTA-456 administration
Time Frame: 48 hours
Population: All patients who received MGTA-456 investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | MGTA-456 Cohort 1 | MGTA-456 Cohort 2
Number analyzed (Participants) | 6 | 2
Participants
  Nausea | 5 | 1
  Hypoalbuminemia | 4 | 1
  Anemia | 4 | 1
  Hypertension | 4 | 1
  Hypocalcemia | 3 | 1
  Leukopenia | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the start of the patient's conditioning regimen (Day -9) up until the patient's 1 year follow-up visit.
Groups:
- MGTA-456: MGTA-456 is an expanded CD34+ cell therapy investigational product used in replacement of single umbilical cord blood transplantation.
  .
Arm/Group | MGTA-456
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MGTA-456 (N=8)
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 3 — Not related to MGTA-456
Immune thrombocytopenia (Blood and lymphatic system disorders) | 3 — Not related to MGTA-456
Pyrexia (General disorders) | 3 — Not related to MGTA-456
Pneumonia (Infections and infestations) | 2 — Not related to MGTA-456
Sepsis (Infections and infestations) | 2 — Not related to MGTA-456
Staphylococcal bacteremia (Infections and infestations) | 2 — Not related to MGTA-456
Autoimmune pancytopenia (Blood and lymphatic system disorders) | 2 — Not related to MGTA-456
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MGTA-456 (N=8)
Anemia (Blood and lymphatic system disorders) | 7 — Not related to MGTA-456
Neutropenia (Blood and lymphatic system disorders) | 7 — Not related to MGTA-456
Thrombocytopenia (Blood and lymphatic system disorders) | 7 — Not related to MGTA-456
Hypertension (Vascular disorders) | 7
Constipation (Gastrointestinal disorders) | 6 — Not related to MGTA-456
Nausea (Gastrointestinal disorders) | 6
Pyrexia (General disorders) | 6 — Not related to MGTA-456
Immune thrombocytopenia (Blood and lymphatic system disorders) | 5 — Not related to MGTA-456
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 — Not related to MGTA-456
Leukopenia (Blood and lymphatic system disorders) | 5 — Not related to MGTA-456

LIMITATIONS AND CAVEATS:
Magenta discontinued the enrollment of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03406962/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03406962/SAP_001.pdf